CLINICAL TRIAL: NCT01653990
Title: A Single-center, Randomized, Double-blinded, 2-way Crossover, Placebo-controlled Study to Assess the QT/QTc Interval After Administration of Single Oral Dose of 400mg Moxifloxacin in Healthy Chinese Subjects
Brief Title: Moxifloxacin_QT Study in Chinese Healthy Volunteer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Haiyan Li, Director of Drug Clinical Trial Center, Peking University Third Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DCTC_2012001
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: QT Interval Prolongation
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- moxifloxacin, pill (Experimental): Oral dose of 400mg moxifloxacin
  Interventions: Drug: moxifloxacin; Drug: moxifloxacin-placebo
- moxifloxacin-placebo,pill (Placebo Comparator): A pill of moxifloxacin-placebo
  Interventions: Drug: moxifloxacin; Drug: moxifloxacin-placebo

INTERVENTIONS:
Drug: moxifloxacin — oral dose of 400mg moxifloxacin
Drug: moxifloxacin-placebo — Oral dose of a pill of moxifloxacin-placebo

SUMMARY:
A single-center, randomized, double-blinded, 2-way crossover, placebo-controlled study to assess the QTc interval after administration of single oral dose of 400mg Moxifloxacin in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese subjects, male, 20 to 45 years of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
2. At Screening, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the subject has rested for 5 minutes. All of vital signs should be within normal ranges:

   * Body temperature (Body) between 35.0-37.0°C
   * 90 ≤ systolic blood pressure <140 mm Hg
   * 60≤ diastolic blood pressure < 90 mm Hg
   * 50≤ pulse rate ≤ 100
3. Body weight need to be at least 50kg or above, 19kg/m2≤ Body Mass Index(BMI) ≤25kg/m2
4. Be able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent prior to any screening procedures.

Exclusion Criteria:

1. History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, genetic or psychiatric disorders.
2. A past medical history of clinically significant ECG abnormalities or a family history (grandparents, parents and siblings) of long QT syndrome, or QTc interval > 440 ms for male or any abnormal ECG findings at screening.
3. Medical histories of syncope, electrophysiological changes, heart failure, reduced exercise tolerance, cardiomyopathy, pericarditis, myocarditis or other cardiac disorders as determined by the investigator.
4. Current electrolyte abnormalities (specifically hypokalemia) in laboratory examination during the screening that are clinical significant as determined by investigator.
5. Current or recent history (< 30 days prior to Screening) of a clinically significant illness.
6. Use of any prescription drugs, herbal supplements, within 4 weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within 4 week prior to initial dosing.
7. Positive results of human immunodeficiency virus, Hepatitis B surface antigen or Hepatitis C antibody testing.
8. History of any hypersensitivity or allergic reaction of moxifloxacin or other types fluoroquinolones.
9. Use of tobacco or history of use of tobacco ( > 5 tobacco/week) or nicotine-containing products in the 3 months prior to screening.
10. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening and/or at baseline.
11. Dosing of study drug in any clinical investigation within 3 months prior to initial dosing.
12. Donation or loss of 200 ml or more of blood within 3 months prior to participation, or donation of component blood within 3 months prior to participation.
13. Consumption of alcohol-, caffeine --containing foods or beverages within 48 hours preceding study drug administration.
14. Other conditions which investigator deems potential harm to subjects if participate the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
baseline-adjusted, placebo-corrected effect on QTcF (ΔΔQTcF) | 1 month

SECONDARY OUTCOMES:
Heart rate, PR, QRS, QTcB and QTcI | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital Drug Clinical Trial Center, Beijing, China